CLINICAL TRIAL: NCT06355622
Title: Pain in RASopathies: New Investigative Techniques and Possible Treatments
Brief Title: Prevalence and Characterization of Pain in RASopathies
Acronym: 3717
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3717
Record Dates: First submitted 2023-02-27; First posted 2024-04-09 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-03

CONDITIONS: RASopathy; Costello Syndrome; Cardio-Facio-Cutaneous Syndrome; Noonan Syndrome
MeSH Terms: conditions — Costello Syndrome; Cardiofaciocutaneous syndrome; Noonan Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case group (Experimental): Detection and characterization of pain by clinical evaluations, biochemical analysis and instrumental tests
  Interventions: Diagnostic Test: Characterization of pain

INTERVENTIONS:
Diagnostic Test: Characterization of pain — Standardized scales and questionnaires to detect and characterize pain, blood sample for pain biomarkers, neurophysiological tests

SUMMARY:
RASopathies are a group of syndromes caused by variants in genes belonging to the RAS/MAPK pathway. Pain is a neglected topic in RASopathies but it is frequently complained by affected individuals.

DETAILED DESCRIPTION:
To detect prevalence and characteristics of pain in RASopathies by using scales, questionnaires, biochemical analysis and neurophysiological assessment tests.

ELIGIBILITY:
Inclusion Criteria:

* All individuals with clinical and molecularly confirmed diagnosis of a RASopathy

Exclusion Criteria:

* Individuals with a RASopathy con confirmed by genetic analysis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pain in verbal patients with RASopathies | 2 years
  To detect the prevalence of pain in verbal patients with RASopathies by using VAS (visual analogue scale) or NRS (numeric rating sclae). Both scales include a range from 0 to 10 where 0 represents no pain, 1-3 range represents mild pain, 4-6 range represents moderate pain and 7-10 range represents severe pain.
Prevalence of Pain in no-communitating patients with RASopathies | 2 years
  To detect the prevalence of pain in no-communicating patients with RASopathies by using FLACC scale. The FLACC Scale includes 5 behavioral categories: facial expression, leg movement, bodily activity, cry or verbalization, and consolability. The parents rated their child's pain at its worst within the preceding 24 h in each category on a scale of 0 to 2, thus an overall pain score ranging from 0 to 10.

SECONDARY OUTCOMES:
Characterization of pain in RASopathies | 2 years
  To detect pain location (one site or multiple body sites) by showing a body map (front and back)

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Leoni, MD, PhD, Principal Investigator — Fondazione Policlinico A. Gemelli, IRCCS
Locations (1):
- Department of Woman and Child Health and Public Health, Fondazione Policlinico A. Gemelli, IRCCS, Roma, Italy